CLINICAL TRIAL: NCT04607889
Title: Measurement of Patient Views on the Attributes of Cancer Genomic Medicine in Japan (Patient View Study)
Brief Title: A Study to Learn More About What Japanese Patients With Solid Tumors Think About Taking Medicine That is Based on Their Genetic Information
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21421
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Cancer Genomic Profiling
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Part 1 - Attribute development: An elicitation phase to develop the list of attributes and levels based on literature review and telephone interviews with patients.
  Interventions: Other: Survey
- Part 2 - Pilot study: A pilot phase consisting of a self-administered, online survey, to be completed by patients and physicians, followed by telephone interviews with a subsample of participants.
  Interventions: Other: Survey
- Part 3 - Main study: The main study, with a self-administered, online survey, to be completed by cancer patients and physicians.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Interviews with study participants will be conducted by telephone or teleconference. The interview will focus on the participants experience with genomic tests, with the expectations, reasons for taking or declining it, hurdles encountered, satisfaction among the key themes to be discussed.
  Other Names: Interviews

SUMMARY:
Researchers are looking for a better way to treat people with solid tumors. One new way is called cancer genomic medicine. In cancer genomic medicine, doctors use tests to look at the genetic information in a solid tumor. These tests are called panel tests. The results of the panel tests help doctors to choose the best type of medicine to treat that tumor.

In this study, the researchers want to learn more about what a large number of patients with solid tumors think are the burden and benefits of taking panel tests. The researchers also want to know what doctors who treat patients with solid tumors think about panel tests.

The study will include about 650 men and women in Japan who are at least 20 years old. About 340 of the participants will be patients with solid tumors who are taking medicine to help treat their tumors. About 310 of the patients will be doctors who are treating patients with solid tumors.

There will be 3 parts in this study. Part 1 will include patients with solid tumors. Parts 2 and 3 will include patients with solid tumors and doctors who are treating patients with solid tumors. In each part, the patients and doctors will answer questions about what they think of panel tests. During Part 1, all of the patients will answer questions in a teleconference. Some of the patients and physicians in Part 2 will also answer questions in a teleconference. During Part 2 and Part 3, all of the patients and doctors will complete an online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Adult female or male patient
* Diagnosis of a solid tumor
* Patients familiar with panel tests to be defined as:

  * Patients who have taken a panel test
  * Patients who have not taken a panel test

    * Patients who have tried or considered taking a panel test
    * Patients who have been offered a panel test but refused
* Signed informed consent
* Is 20 years of age or older

Part 2 and Part 3 (patients):

* Female or male patient
* Diagnosis of a solid tumor (lung, or one of rare tumors defined by National Cancer Center and MHLW: mouth and lip, ovary and fallopian tube, urinary tract, soft tissue sarcoma, neuroendocrine, glioma, oropharynx, salivary, testis, parathesis, teratoma, skin melanoma, small intestine, nasal, nasal sinus, skin appendages, mesothelioma, GIST, vaginal and vulvar, thymic, nasopharynx, bone sarcoma, anus, uterine carcinosarcoma, penile, extragonadal germ cell, embryonal carcinoma, mucosa melanoma, pineal, brain and CNS, eye, peripheral nerve, trachea, melanoma of uvea, meningioma, histocytic and dendritic cell, trophoblastic tumor of placenta, Kaposi sarcoma, middle ear)
* Sees the doctor for cancer treatment on regular basis (at least once every three months)
* Signed informed consent
* Is 20 years of age or older

Part 2 and Part 3 (physician):

* Has prescribed anti-cancer drugs to patients with a solid tumor (lung or one of rare tumors defined by National Cancer Center and MHLW: mouth and lip, ovary and fallopian tube, urinary tract, soft tissue sarcoma, neuroendocrine, glioma, oropharynx, salivary, testis, parathesis, teratoma, skin melanoma, small intestine, nasal, nasal sinus, skin appendages, mesothelioma, GIST, vaginal and vulvar, thymic, nasopharynx, bone sarcoma, anus, uterine carcinosarcoma, penile, extragonadal germ cell, embryonal carcinoma, mucosa melanoma, pineal, brain and CNS, eye, peripheral nerve, trachea, melanoma of uvea, meningioma, histocytic and dendritic cell, trophoblastic tumor of placenta, Kaposi sarcoma, middle ear) in the last 3 months.
* Signed informed consent

Exclusion Criteria:

Part 1:

* Non-Japanese speakers
* Declaring to be too unwell to perform an interview

Part2 and Part 3 (patients):

* Non-Japanese speakers
* Declaring to be too unwell to complete the survey
* Participation in the pilot study

Part 2 and Part 3 (physician):

- Non-Japanese speakers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Part 1:
  Adult female and male patients with a diagnosis of a solid tumor, who have taken or tried to take a panel test will be enrolled in the study.
  Part 2 and Part 3 (patients):
  Female and male patients with a diagnosis of a solid tumor and will be enrolled in the study.
  Part 2 and Part 3 (physicians):
  Physicians with experience in genomic medicine will be preferred as study participants but the sample will not be limited to them.
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Best-Worst Scaling scores showing patient preferences for the attributes of the process of taking panel tests | Up to 25 minutes
  Respondents will choose "Best" or "Worst" for prepared questions.

SECONDARY OUTCOMES:
Best-Worst Scaling scores showing doctor preferences for the attributes of the process of taking panel tests | Up to 25 minutes
  Doctors will choose "Best" or "Worst" for prepared questions.
Ranking of Best-Worst scaling scores for patients and for doctors | Up to 25 minutes
  Attributes will be ranked based on the responses by patients and doctors.
Patient and doctor willingness to try/offer panel tests based on different hypothetical conditions of panel tests and drugs in cancer genomic medicine | Up to 25 minutes
  Willingness to try questions based on hypothetical conditions would enable the policy makers and thought leaders improve the clinical practice of cancer genomic medicine in a patient-centric way.

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Suehara Y, Hasegawa K, Majima Y, Mita N, Barbier S, Bogoeva N, Kato S. Patient and physician preferences for cancer panel testing in Japan: a best-worst scaling study. BMJ Open. 2025 Aug 26;15(8):e097620. doi: 10.1136/bmjopen-2024-097620. PMID 40858382